CLINICAL TRIAL: NCT05953870
Title: Music Therapy to Reduce Perioperative Stress and Increase Satisfaction in Patients Undergoing Ambulatory Surgery: a Randomized Trial
Brief Title: This is a Study to Evaluate if Music Therapy Can Reduce Stress and Increase Satisfaction of Patients Undergoing Ambulatory Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORBV-CHIR-003
Record Dates: First submitted 2023-06-23; First posted 2023-07-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Stress; Personal Satisfaction
MeSH Terms: conditions — Personal Satisfaction | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUSIC AND COMFORT THERAPY (Experimental): The intervention group will be "exposed" pre- and postoperatively to relaxing music, which is defined as a slower tempo music that can quiet mind and make patients feel soothed.
  Interventions: Other: Music Therapy
- CONTROL GROUP (No Intervention): These patients will follow the standard surgical pathways as per daily routine.

INTERVENTIONS:
Other: Music Therapy — slower tempo music that can quiet mind and make patients feel soothed
  Arms: MUSIC AND COMFORT THERAPY

SUMMARY:
Patients who undergo outpatient surgery according to normal practice will be divided into two groups.

The first group (17 patients), before and after their surgery, will listen to relaxing music, namely a slower tempo music that can quiet mind and make patients feel soothed.

The second group (17 patients) will follow the standard surgical pathways according to normal clinical practice, in particular they will not listen to relaxing music.

A questionnaire to evaluate stress and satisfaction will be administered to all the patients before their discharge

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing outpatient surgery
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Concern | during hospitalization, 1 day
  Concern (measured on the validated Leiden Perioperative Patient Satisfaction -LPPS - questionnaire for the perioperative patients' satisfaction). This questionnaire assess patient satisfaction with perioperative care. Patients are asked to score each question on a fivepoint scale (from 1 - corresponding to the worse outcome to 5 - the best outcome)

SECONDARY OUTCOMES:
Personal satisfaction | during hospitalization, 1 day
  In hospital satisfaction (measured on the validated Leiden Perioperative Patient Satisfaction -LPPS - questionnaire for the perioperative patients' satisfaction. This questionnaire assess patient satisfaction with perioperative care. Patients are asked to score each question on a fivepoint scale (from 1 - corresponding to the worse outcome to 5 - the best outcome)
Length of hospital stay | during hospitalization, 1 day
  number of hours the participant is being hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Davide La Regina, MD, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Ospedale Regionale Bellinzona e Valli, Ente Ospedaliero Cantonale, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided